CLINICAL TRIAL: NCT04987203
Title: TiNivo-2: A Phase 3, Randomized, Controlled, Multicenter, Open-label Study to Compare Tivozanib in Combination With Nivolumab to Tivozanib Monotherapy in Subjects With Renal Cell Carcinoma Who Have Progressed Following One or Two Lines of Therapy Where One Line Has an Immune Checkpoint Inhibitor
Brief Title: Study to Compare Tivozanib in Combination With Nivolumab to Tivozanib Monotherapy in Subjects With Renal Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AVEO Pharmaceuticals, Inc. (Industry)
Collaborators: Parexel (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AV-951-20-304
Record Dates: First submitted 2021-07-23; First posted 2021-08-03 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Renal Cell Carcinoma
Keywords: Immune Checkpoint Inhibitor; Open-label; Monotherapy; Disease Progression
MeSH Terms: conditions — Carcinoma, Renal Cell; Disease Progression | interventions — tivozanib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tivozanib in Combination with Nivolumab (Experimental): Subjects with advanced RCC will receive 0.89 mg of tivozanib once daily (QD) for 3 weeks followed by 1 week off study drug and nivolumab every 4 weeks on Day 1 of each Cycle, until disease progression or unacceptable toxicities occur, other withdrawal criteria are met, or completion of 2 years of treatment [for nivolumab] whichever occurs first.
  Interventions: Drug: Tivozanib; Drug: Nivolumab
- Tivozanib (Experimental): Subjects with advanced RCC will receive 1.34 mg of tivozanib once daily (QD) for 3 weeks followed by 1 week off study drug until disease progression or unacceptable toxicities occur, or other withdrawal criteria are met.
  Interventions: Drug: Tivozanib

INTERVENTIONS:
Drug: Tivozanib — Tivozanib will be administered orally.
Drug: Nivolumab — Nivolumab will be administered via intravenous infusion.
  Arms: Tivozanib in Combination with Nivolumab

SUMMARY:
This study will be comparing tivozanib in combination with nivolumab to tivozanib alone in subjects with advanced Renal Cell Carcinoma (RCC) who have had 1 or 2 prior lines of therapy, one of which was an Immune Checkpoint Inhibitor (ICI).

DETAILED DESCRIPTION:
This will be an open-label, randomized, controlled, multicenter, multi-national, parallel-arm study. The study is designed to compare the progression free survival (PFS), overall survival (OS), Objective response rate (ORR), duration of response (DoR), and safety of tivozanib and the combination of tivozanib with nivolumab.

Approximately 326 subjects with refractory advanced RCC at approximately 190 sites will be randomized in a 1:1 ratio to treatment with tivozanib plus nivolumab (163 subjects) or tivozanib (163 subjects). Subjects will be randomly assigned to a treatment.

Subjects will receive 1.34 mg/day (monotherapy arm) or 0.89mg/day (combination arm) of tivozanib once daily (QD) for 3 weeks followed by 1 week off study drug. One cycle will be defined as 4 weeks: 3 weeks on treatment and 1 week off treatment. Subjects who receive nivolumab will be infused with 1 treatment of nivolumab at specified dose on specified days of each Cycle.

Subjects with documented stable disease or an objective response may continue to receive both tivozanib and nivolumab therapy at the same dose and schedule until progression as long as the tolerability is acceptable. Nivolumab will be discontinued in all subjects after 2 years; Tivozanib may be continued after discontinuation of nivolumab until other withdrawal criteria are met. A Safety Follow-up Visit will be performed 30 days (± 7 days) after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Radiographic disease progression during or following at least 6 weeks of treatment with ICI for locally advanced or metastatic RCC with a clear cell component either in first- or second-line treatment.
* Subjects must have recovered from the adverse events of prior therapy to grade ≤ 1 or baseline.
* Histologically or cytologically confirmed RCC with a clear cell component.
* Measurable disease per RECIST criteria Version 1.1.
* Eastern Cooperative Oncology Group performance status of 0 or 1.
* All participants must follow protocol defined contraceptive measures.

Exclusion Criteria:

* Subjects who received: a. A single agent tyrosine kinase inhibitor (TKI) in the first line setting followed by a single agent immune checkpoint inhibitor (ICI) in the second line setting; b. More than 2 prior lines of therapy in the advanced or metastatic setting.
* History of life-threatening toxicity related to prior immune therapy.
* Active autoimmune disease as well as those that required discontinuation of prior immuno-oncological (IO) therapy due to immune mediated AEs.
* Uncontrolled hypertension.
* More than 1 prior line of therapy with a checkpoint inhibitor in the metastatic setting.
* Subjects on immune suppressive therapy for organ transplant or subjects with a history of genetic or acquired immune suppression disease such as human immunodeficiency virus (HIV) [Patients with HIV who have CD4+ T-cell counts >350 cells/µL, without a history of acquired immune deficiency syndrome (AIDS)-defining opportunistic infections, and are on established antiretroviral therapy which does not include a cytochrome P450 (CYP)3A4 inducer, for at least 4 weeks and have an HIV viral load less than 400 copies/mL, are eligible].
* History of clinically significant interstitial lung disease or current non-infectious pneumonitis.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | Until progressive disease [PD] (Approximately 30 months)
  Comparison of the PFS of tivozanib in combination with nivolumab to tivozanib in subjects with RCC who have progressed following 1 or 2 lines of therapy. PFS is defined as the time from randomization to first documentation of objective tumor progression (progressive disease [PD], radiological) according to Response Evaluation Criteria In Solid Tumors (RECIST), or death due to any reasons whichever comes first.

SECONDARY OUTCOMES:
Overall Survival | From Screening (Days -28 to -1) until death (Approximately 42 months)
  Comparsion of the OS of subjects randomized to treatment with tivozanib in combination with nivolumab compared to tivozanib. OS is defined as the time from the date of randomization to date of death due to any cause.
Progression free survival | Until progressive disease [PD] (Approximately 30 months)
  PFS is defined as the time from randomization to first documentation of objective tumor progression (progressive disease [PD], radiological) according to RECIST, or death due to any reasons whichever comes first. PFS as assessed by investigator.
Objective Response Rate | From Screening (Days -28 to -1) until PD (Approximately 30 months)
  Comparison of ORR of subjects randomized to treatment with tivozanib in combination with nivolumab compared to tivozanib. ORR is defined as the proportion of subjects with confirmed complete response or confirmed partial response according to RECIST relative to the total population of randomized subjects.
Duration of Response | From Screening (Days -28 to -1) until PD or death (Approximately 30 months)
  Comparison of DoR of subjects randomized to treatment with tivozanib in combination with nivolumab compared to tivozanib. DoR is defined as the time from the first documentation of objective tumor response to the first documentation of objective tumor progression or to death due to any cause.
Number of subjects with serious and non-serious adverse events | From Screening (Day -28 to Day -1) to Follow-up visit (30 days after last dose of study drug ± 7 days)
  Assessment of the safety and tolerability of tivozanib in combination with nivolumab compared to tivozanib.

CONTACTS AND LOCATIONS:
Locations (139):
- United States (36):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Chao Family Comprehensive Cancer Center, UC Irvine, Irvine, California
  - University of California San Diego, La Jolla, California
  - Leland Stanford Junior University, Redwood City, California
  - Kaiser Permanente Riverside Medical Center, Riverside, California
  - US Oncology - Rocky Mountain Cancer Centers - Midtown, Denver, Colorado
  - Florida Cancer Specialists & Res Inst, Fort Myers, Florida
  - Florida Cancer Specialists & Research Institute (FCS) - Tampa Cancer Center Location, St. Petersburg, Florida
  - The University of Kansas Cancer Center, Westwood, Kansas
  - University of Kentucky UK Markey Cancer Center, Lexington, Kentucky
  - Tulane Cancer Center Clinic - Oncology, New Orleans, Louisiana
  - University of Maryland Medical Center-Greenebaum Cancer Ctr, Baltimore, Maryland
  - John Hopkins Medicine - Hematology/oncology, Baltimore, Maryland
  - Maryland Oncology Hematology, Clinton, Maryland
  - Dana-Farber Cancer Institute - Medicine, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - St. Vincent Frontier Cancer Center, Billings, Montana
  - Oncology Hematology West PC dba Nebraska Cancer Specialists, Omaha, Nebraska
  - Memorial Sloan Kettering Cancer Center - Monmouth - Oncology, Middletown, New Jersey
  - University of New Mexico - Comprehensive Cancer Center, Albuquerque, New Mexico
  - Roswell - Roswell Park Cancer Institute - Medical Oncology, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center - Westchester, East White Plains, New York
  - Memorial Sloan Kettering Cancer Center (MSKCC) - Memorial Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center - Nassau, Uniondale, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Lehigh Valley Physician Group, Allentown, Pennsylvania
  - Allegheny General Hospital (AGH), Pittsburgh, Pennsylvania
  - UH Cleveland Medical Center, Columbia, South Carolina
  - Chattanooga Oncology and Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Oncology - Central Austin Cancer Center, Austin, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - US Oncology Texas Oncology (CCC of South Texas) - San Antonio Medical Center, San Antonio, Texas
  - University Of Washington - Medical Center, Seattle, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
- Argentina (4):
  - Centro Oncológico Korben, Buenos Aires, Ciudad Autónoma de Buenos Aire
  - Clínica Viedma, Viedma, Río Negro Province
  - Centro Oncologico de Rosario, Rosario, Santa Fe Province
  - Centro para la Atención Integral del paciente Oncológico, San Miguel de Tucumán, Tucumán Province
- Australia (4):
  - Liverpool Hospital Cancer Therapy Centre, Liverpool, New South Wales
  - Mater Misericordiae Limited, Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Sunshine Hospital, Geelong, Victoria
- Belgium (6):
  - ZNA Jan Palfijn, Merksen, Antwerpen
  - Institut Jules Bordet - Oncologie Médicale, Anderlecht, Brussels Capital
  - Jessa Ziekenhuis - Campus Virga Jesse - Medische Oncologie, Hasselt, Limburg
  - UZ Gent - Medische Oncologie, Ghent, Oost-Vlaanderen
  - CHU Brugmann - Victor Horta, Brussels
  - AZ Groeninge - Campus Kennedylaan, Kortrijk
- Brazil (6):
  - Centro Gaucho Integrado de Onc, Porto Alegre, Rio Grande do Sul
  - Clinica de Neoplasias Litoral, Itajaí, Santa Catarina
  - Universidade Estadual de Campi, Campinas, São Paulo
  - Instituto Brasileiro de Controle do Cancer - ibcc, São Paulo, São Paulo
  - Hospital Nossa Senhora da Conc, Porto Alegre
  - Pontificia Universidade, Porto Alegre
- Canada (4):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - BC Cancer - Vancouver Centre, Vancouver, British Columbia
  - Sunnybrook Research Institute, sunnybrook Health Sciences Ct, Toronto, Ontario
  - University Health Network - Princess Margaret Cancer Centre, Toronto, Ontario
- Chile (4):
  - ACEREY Centro de Investigación Clínica Oncológica, Viña del Mar, Región de Valparaíso
  - Centro de Estudios Clinicos In, Santiago, Región Metropolitana de Santia
  - Centro de Estudios Clínicos SAGA SpA, Santiago, Región Metropolitana de Santia
  - Meditek Ltda., Santiago, Santiago Metropolitan
- Czechia (4):
  - University Hospital Brno, Brno, Brno-město
  - Fakultni Thomayerova nemocnice, Prague, Praha 4
  - FN Hradec Kralove, Hradec Králové
  - FN Kralovske Vinohrady, Prague
- France (16):
  - Institut de cancérologie de Strasbourg Europe - ICANS, Strasbourg, Alsace
  - Hospices Civils de Lyon (HCL) - Centre Hospitalier Lyon-Sud, Pierre-Bénite, Auvergne-Rhône-Alpes
  - Institut Paoli Calmettes - HÃ´pital de jour, Marseille, Bouches-du-Rhône
  - Hopital Saint-Andre - Service d'Oncologie Medicale, Bordeaux, Gironde
  - Hopital Foch, Suresnes, Hauts-de-Seine
  - CHU Michallon - Hopital Nord - Cancérologie Et Hématologie, Grenoble, Isère
  - Hôpital privé Le Bois, Lille, Nord
  - Centre Hospitalier de Poitiers, Poitiers, Poitou-Charentes
  - Centre Leon Berard - departement d'oncologie medicale, Lyon, Rhône
  - Clinique Victor Hugo - Hematologie, Le Mans, Sarthe
  - CHD Vendee La Roche sur Yon - Gastro-Entérologie, La Roche-sur-Yon
  - Centre de Lutte Contre le Cancer (CLCC), Nice
  - ICO - Site Rene Gauducheau - Oncologie Medicale, Saint-Herblain
  - Hopital Trousseau - medical oncology, Tours
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Centre de Lutte Contre le Cancer (CLCC) - Gustave Roussy (Institut de Cancerologie Gustave-Roussy), Villejuif, Île-de-France Region
- Germany (2):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
- Italy (12):
  - Ospedale S.Donato, AUSL 8 di Arezzo, Arezzo, Arezzo
  - Azienda Mater Domini, Catanzaro, Catanzaro
  - P.O. Ss. Annunziata, Chieti Scalo, Chieti
  - IRST, Meldola (Fc), Forli
  - European Institute of Oncology, Milan, Milano
  - IRCCS Policlinico San Matteo, Pavia, Pavia
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma, Roma
  - AO S.Camillo-Forlanini, Roma, Roma
  - Azienda Ospedaliera Santa Maria di Terni, Terni, Terni
  - PO di Cremona, ASST di Cremona - Oncologia medica, Cremona
  - AOUC Azienda Ospedaliero-Universitaria Careggi, Florence
  - IRCCS Fondazione "Giovanni Pas, Napoli
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Tlalpan, Mexico
- Poland (9):
  - Szpital Kliniczny Przemienienia Panskiego UM w Poznaniu, Poznan, Greater Poland Voivodeship
  - Szpital Specjalistyczny im. L. Rydygiera w Krakowie, Krakow, Lesser Poland Voivodeship
  - Europejskie Centrum Zdrowia Otwock, Szpital im. F. Chopina, Otwock, Masovian Voivodeship
  - Szpital Specjalist. w Brzozowie,Podkarpacki Ośrodek Onkologi, Brzozów, Podkarpackie Voivodeship
  - Nzoz Mrukmed Lekarz Beata Madej-Mruk I Partner Sp. P., Rzeszów, Podkarpackie Voivodeship
  - COPERNICUS Podmiot Leczn. Sp z o.o.,Wojew. Centrum Onkologii, Gdansk, Pomeranian Voivodeship
  - Wojewodzki Szpital Specjalistyczny, Biała Podlaska
  - Centralny Szpital Kliniczny Ministerstwa Spraw Wewnetrznych, Warsaw
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie - Państwowy Instytut Badawczy, Warsaw
- Portugal (5):
  - Hospital Particular do Algarve - Gambelas-Faro, Faro, Faro District
  - H. Prof. Doutor Fernando Fonseca, Amadora, Lisbon District
  - H. de Santa Maria. Centro Hospitalar Lisboa Norte - Oncologia, Lisbon, Lisbon District
  - H. Santo Antonio. Centro Hospitalar do Porto, Porto, Porto District
  - Instituto Português Oncologia Francisco Gentil do Porto, Porto
- Spain (16):
  - H.G.U. de Elche, Elche, Alicante
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital de La Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Universitario Vall d', Barcelona, Barcelona
  - Institut Catalá d´Oncología (I.C.O.), Barcelona, Barcelona
  - Hospital Del Mar, Barcelona, Barcelona
  - Hospital Universitari Parc Tau, Sabadell, Barcelona
  - ICO-Hospital Universitari de G, Girona, Girona
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital U. 12 Octubre, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Universitario Virgen, Seville, Sevilla
  - Fundación Instituto Valenciano, Valencia, Valencia
  - Hospital Universitario Y Politécnico La Fe, Valencia, Valenciana, Comunidad
  - C.H.U. de Orense, Ourense
- United Kingdom (10):
  - Addenbrooke's Hospital - Oncology, Cambridge, Cambridgeshire
  - Mount Vernon Cancer Centre, Northwood, England
  - Royal Blackburn Hospital - Oncology, Preston, Lancashire
  - Imperial College Healthcare NHS Trust - Hammersmith Hospital, London, London, City of
  - The Christie NHS Foundation Trust - Medical Oncology, Manchester, Manchester
  - Royal Marsden - Sutton, Sutton, Surrey
  - Royal Marsden Hospital, Sutton, Surrey
  - New Cross Hospital, Wolverhampton, Wolverhampton
  - Royal Derby Hospital, Derby
  - Leeds Teaching Hospitals NHS Trust, Leeds

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choueiri TK, Albiges L, Barthelemy P, Iacovelli R, Emambux S, Molina-Cerrillo J, Garmezy B, Barata P, Basu A, Bourlon MT, Moon H, Ratta R, McKay RR, Chehrazi-Raffle A, Hammers H, Heng DYC, Braendle E, Beckermann KE, McGregor BA, Motzer RJ. Tivozanib plus nivolumab versus tivozanib monotherapy in patients with renal cell carcinoma following an immune checkpoint inhibitor: results of the phase 3 TiNivo-2 Study. Lancet. 2024 Oct 5;404(10460):1309-1320. doi: 10.1016/S0140-6736(24)01758-6. Epub 2024 Sep 13. PMID 39284329
- [Derived] Yang Y, Psutka SP, Parikh AB, Li M, Collier K, Miah A, Mori SV, Hinkley M, Tykodi SS, Hall E, Thompson JA, Yin M. Combining immune checkpoint inhibition plus tyrosine kinase inhibition as first and subsequent treatments for metastatic renal cell carcinoma. Cancer Med. 2022 Aug;11(16):3106-3114. doi: 10.1002/cam4.4679. Epub 2022 Mar 18. PMID 35304832